CLINICAL TRIAL: NCT02700594
Title: Effect of Hip Versus Spinal Joint Mobilization on Hip Muscle Strength
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S13-00683
Record Dates: First submitted 2014-09-23; First posted 2016-03-07 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-03

CONDITIONS: Joint; Derangement, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hip mobilization (Active Comparator): Prone posterior-to-anterior Grade IV hip joint mobilization: The subject will be placed in prone on a treatment table. The intervening physical therapist will place the heel of his hand on the greater trochanter of the femur on the involved side provide rhythmic anterior-directed force. The subject will receive 3 bouts of 30 seconds of continuous mobilizations with 10 seconds rest in between bouts. For the prone posterior-to-anterior Grade IV hip joint mobilization, the intervening therapist will perform all 3 bouts in the same position.
  Interventions: Other: Joint mobilization
- Spine mobilization (Active Comparator): Prone unilateral posterior-to-anterior Grade IV lumbar spinal joint mobilization: The subject will be placed in prone on the treatment table. The intervening physical therapist will place his thumbs on the transverse process, on the affected side, of the L3, L4 or L5 vertebrae and provide a rhythmic anterior-directed force. Prone unilateral posterior-to-anterior Grade IV lumbar spinal joint mobilization, the intervening therapist will perform 1 bout on each of L3, L4 and L5 for a total of 3 bouts
  Interventions: Other: Joint mobilization

INTERVENTIONS:
Other: Joint mobilization — Mobilization and manipulation are manual therapy techniques" comprising a continuum of skilled passive movements to the joints and/or related soft tissues that are applied at varying speeds and amplitudes, including a small-amplitude/high- velocity therapeutic movement."16 The term joint mobilization, or nonthrust mobilization, often refers to slow, "rhythmic, repetitive passive movements to the patients' tolerance, in voluntary and/or accessory range and graded according to examination findings."

SUMMARY:
Patients with painful knee conditions often present with hip muscle weakness. This weakness can lead to, and perpetuate, knee problems. Diminished strength causes movement impairments that can lead to pathology, functional limitations and disablement. In some cases, this hip muscle weakness is not caused by simple disuse and muscle shrinkage (atrophy). Hip weakness may be caused by an inhibitory mechanism that limits the force output of a muscle. The inhibition is reflexive and is in response to pain or joint dysfunction. Joint mobilization/manipulation can quickly reduce pain and improve joint function, possibly decreasing inhibition and increasing strength. Joint mobilization/manipulation may facilitate strength recovery. By restoring strength sooner, the patient may avoid the deleterious effects of prolonged muscle weakness and achieve quicker or better outcomes.

DETAILED DESCRIPTION:
Patients with knee pain often present with hip muscle weakness. Hip muscle weakness can cause faulty hip mechanics that contribute to adverse knee joint kinematics. The gluteus maximus is the largest hip muscle and its primary actions are extension and external rotation of the hip joint. Gluteus muscle weakness was associated with varied knee injuries, including patellofemoral pain syndrome, iliotibial band syndrome and anterior cruciate ligament (ACL) sprains. In 2 systematic reviews that have assessed subjects with anterior knee pain, the authors found strong evidence for impaired hip extensor muscle strength and activation. In a prospective cohort study, weak hip external rotation strength was associated with the development of anterior knee pain and the hip strength further diminished after pain started. There is evidence supporting gluteal muscle strengthening for the management of anterior knee pain. Some authors argue that gluteal muscle weakness may be caused by muscle inhibition and not simple disuse atrophy. This reflexive muscle inhibition is neural-mediated and driven by pain or joint dysfunction. Joint mobilization/manipulation reduces pain and improves joint function and may help maximize strength by reducing inhibition. Yerys et. al. (2002) demonstrated that hip joint mobilization caused an immediate 14% increase gluteus maximus strength and Makofsky (2007) found an immediate 17% increase in gluteus medius strength after hip joint mobilization. Both of these studies, however, used asymptomatic subjects and their results may not translate to symptomatic patients. Chilibeck (2011) found an immediate 14% increase in hip extension strength, and 12% in hip abduction, after lumbar spine thrust joint manipulation. This study also used an asymptomatic sample. In addition, thrust joint manipulation is used less frequently in physical therapy practice compared to nonthrust joint mobilization. The scientific objective for this research is to assess the effect of spine and hip joint mobilization on hip muscle strength in patients with knee pain.

The study aims to answers the following questions:

1. Does hip joint mobilization immediately improve hip muscle strength in patients with knee pain?
2. Does spinal joint mobilization immediately improve hip muscle strength in patients with knee pain?
3. Does hip or spinal joint mobilization create a greater improvement on hip muscle strength in patients with knee pain?

This pilot, prospective clinical trial will use a randomized clinical trial design. The primary dependent variable is isometric muscle strength, measured in pounds, an interval level of measurement. Muscle strength will be determined by the maximum voluntary contraction (MVC) and measured by an electronic hand-held dynamometer. Hand-held dynamometric muscle testing has demonstrated good intrarater reliability and validity when compared to Biodex dynamometry. Although there is no established minimal clinically important change (MCID) score for strength testing, some authors have suggested a 10% change in strength to be clinically significant. Pain will be measured at the ordinal level with the numeric pain rating scale (NRPS). Investigators will recruit subjects from routine clinical practice within the NYULMC-CMC. The outcomes variables (isometric muscle strength and strength) will be measured before and after the intervention at the initial evaluation visit. After these measures are obtained, the participation in the study is complete. There is no follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Age18-75
2. Referred to out-patient physical therapy for evaluation/treatment of a knee condition
3. Agreed to be in the study and signed the informed consent document

Exclusion Criteria:

1. Presence of any medical 'red flags' suggestive of pain that is not of musculoskeletal origin
2. Osteoporosis or recent fracture of the hip or spinal joints
3. Spinal or hip joint surgery or prosthesis
4. Spinal instability (Grade II spondylolithesis or greater), spondyloarthritides, or severe spinal misalignment
5. Nervous system disease or disorder
6. Pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change in strength from baseline to immediately after intervention (maximum voluntary contraction (MVC) and measured by an electronic hand-held dynamometer) | 1 Hour
  The primary dependent variable is the isometric muscle strength, measured in pounds, an interval level of measurement. Muscle strength will be determined by the maximum voluntary contraction (MVC) and measured by an electronic hand-held dynamometer

SECONDARY OUTCOMES:
Change in pain from baseline to immediately after intervention (numeric pain rating scale (NRPS) | 1 Hour
  Pain will be measured at the ordinal level with the numeric pain rating scale (NRPS

CONTACTS AND LOCATIONS:
Overall Officials: Angela Stolfi, DPT, Principal Investigator — Rusk PT Director

REFERENCES:
- [Background] Bialosky JE, Bishop MD, Price DD, Robinson ME, George SZ. The mechanisms of manual therapy in the treatment of musculoskeletal pain: a comprehensive model. Man Ther. 2009 Oct;14(5):531-8. doi: 10.1016/j.math.2008.09.001. Epub 2008 Nov 21. PMID 19027342
- [Background] Makofsky H, Panicker S, Abbruzzese J, Aridas C, Camp M, Drakes J, Franco C, Sileo R. Immediate Effect of Grade IV Inferior Hip Joint Mobilization on Hip Abductor Torque: A Pilot Study. J Man Manip Ther. 2007;15(2):103-10. doi: 10.1179/106698107790819927. PMID 19066650